CLINICAL TRIAL: NCT01683331
Title: A Clinical Trial to Prevent New Onset Diabetes After Transplantation
Acronym: ITP-NODAT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Akinlolu Ojo, Emeritus Professor of Medicine, Active, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R01DK092475-01 (NIH)
Record Dates: First submitted 2012-08-30; First posted 2012-09-11 (Estimated); Results first posted 2019-03-20 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-02

CONDITIONS: Prevention of New Onset Diabetes Among Kidney Transplant Patients
Keywords: Kidney transplant; New onset diabetes; Prevention; Insulin
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- Insulin treatment for hyperglycemia (Active Comparator): Neutral Protamine Hagedorn (NPH) Insulin Titration Regimen, based on pre-dinner capillary blood glucose measurements (CPG) expressed in mg/dl; All NPH initiation doses and dose adjustments are presented in IU/day For pts. with CPG > 240, NPH initiation: 14, dose increases by 4; For pts. with CPG > 180 mg/dl, NPH initiation: 12, dose increases by 4; For pts. with CPG > 140 mg/dl, NPH initiation: 10, dose increases by 4; For pts. with CPG > 120 mg/dl, NPH initiation: 0, dose increases by 2; For pts. with CPG 100-119 mg/dl, NPH initiation: 0, maintain dose; For pts. with CPG 80-<100 mg/dl, NPH initiation: 0, dose decrease by 4; For pts. with CPG 60-<80 mg/dl, NPH initiation: 0, decrease by 8; For pts. with CPG <60 mg/dl, NPH initiation: 0, ½ of previous dose.
  Interventions: Drug: Insulin treatment for hyperglycemia
- Standard of care (No Intervention): Patients assigned in this arm will receive standard of care following their kidney transplantation.

INTERVENTIONS:
Drug: Insulin treatment for hyperglycemia
  Arms: Insulin treatment for hyperglycemia

SUMMARY:
Specific Aim 1: To determine the clinical efficacy of early initiation of insulin therapy in decreasing the incidence of NODAT among de novo kidney transplant patients with manifested post-transplant hyperglycemia during the first week after transplantation.

Hypothesis 1: Early initiation of insulin therapy protects beta-cell from early stress related to the surgery and use of higher doses of immunosuppressive medications, and leads to lower incidence of NODAT at 1 and 2 years.

Specific Aim 2: To determine the improvement in overall glycemic control with the early initiation of insulin therapy.

Hypothesis 2: Early initiation of insulin therapy results in greater overall control of glycemia compared to standard care of dietary counseling, life-style modification, oral hypoglycemic agents and/or insulin as needed at 1 year.

Specific Aim 3: To determine the improvement in beta-cell function among patients assigned to the early initiation of insulin therapy at one year post-transplantation.

Hypothesis 3: Early initiation of insulin therapy protects beta-cell from glucotoxicity of post-transplant hyperglycemia and preserves better beta-cell function at 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (> 18 years) with end stage renal disease (ESRD) undergoing kidney transplantation;
2. Standard triple immunosuppressive medications following kidney transplantation including tacrolimus, mycophenolate mofetil and corticosteroids;
3. Capable to understand the study protocol and to give informed consent;

Exclusion Criteria:

1. Type 1 and 2 Diabetes Mellitus (DM) either as co-morbidity or cause of ESRD;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2018-02-27 (Actual); Study Completion 2018-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Akinlolu Ojo, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 42 participants randomized prior to kidney transplantation at University of Michigan, 6 did not undergo study procedure due to medical conditions that developed in the immediate postoperative period which prevented them from going forward in the study. Data are not available on the 209 participants randomized through the University of Austria.
Groups:
- Insulin Treatment for Hyperglycemia: NPH Insulin Titration Regimen, based on pre-dinner capillary blood glucose measurements (CPG) expressed in mg/dl; All NPH initiation doses and dose adjustments are presented in IU/day For pts. with CPG > 240, NPH initiation: 14, dose increases by 4; For pts. with CPG > 180 mg/dl, NPH initiation: 12, dose increases by 4; For pts. with CPG > 140 mg/dl, NPH initiation: 10, dose increases by 4; For pts. with CPG > 120 mg/dl, NPH initiation: 0, dose increases by 2; For pts. with CPG 100-119 mg/dl, NPH initiation: 0, maintain dose; For pts. with CPG 80-<100 mg/dl, NPH initiation: 0, dose decrease by 4; For pts. with CPG 60-<80 mg/dl, NPH initiation: 0, decrease by 8; For pts. with CPG <60 mg/dl, NPH initiation: 0, ½ of previous dose.
Period: Overall Study
Arm/Group | Insulin Treatment for Hyperglycemia | Standard of Care
Started | 18 | 18
Began Dosage | 18 | 18
12 Months | 18 | 18
24 Months | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin Treatment for Hyperglycemia | Standard of Care | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.6 (13.9) | 44.6 (15.5) | 48.6 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 8 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 17 | 16 | 33
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 1 | 6
  White | 13 | 16 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: The Incidence of New Onset of Diabetes After Transplant (NODAT) 12 Months After Kidney Transplantation
Description: NODAT will be defined according to American Diabetes Association definition:
  1. Fasting glucose level equal or greater than 126 mg/dl on two separate blood testings; and/or
  2. 2 hours Oral Glucose Tolerance Test (OGTT) values equal or greater than 200 mg/dl; and/or
  3. Glycosylated hemoglobin A1c equal or greater than 6.5; and/or
  4. On oral hypoglycemic agents and/or insulin therapy; Incidence is measured in terms of number of participants who meet any of these 4 criteria.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Treatment for Hyperglycemia | Standard of Care
Number analyzed (Participants) | 18 | 18
Participants | 3 | 1
Statistical Analysis 1: Comparison: Insulin Treatment for Hyperglycemia vs Standard of Care; Test type: Superiority; p = 0.87, Chi-squared; Odds Ratio (OR) = 1.03, 95% CI 2-sided [1.01 to 1.06]

2. Secondary Outcome: The Incidence of New Onset of Diabetes After Transplant (NODAT) 24 Months After Kidney Transplantation
Description: NODAT will be defined according to American Diabetes Association definition:
  1. Fasting glucose level equal or greater than 126 mg/dl on two separate blood testings; and/or
  2. 2 hours OGTT values equal or greater than 200 mg/dl; and/or
  3. Glycosylated hemoglobin A1c equal or greater than 6.5; and/or
  4. On oral hypoglycemic agents and/or insulin therapy;
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Treatment for Hyperglycemia | Standard of Care
Number analyzed (Participants) | 18 | 18
Participants | 1 | 0
Statistical Analysis 1: Comparison: Insulin Treatment for Hyperglycemia vs Standard of Care; Test type: Superiority; p = 0.92, Chi-squared; Odds Ratio (OR) = 1.3, 95% CI 2-sided [1.2 to 2.8]

3. Other Pre Specified Outcome: Incidence of Impaired Fasting Glycemia and Impaired Glucose Tolerance 6, 12 and 24 Months After Transplantation.
Description: Following American Diabetes Association's definition:
  Impaired fasting glycemia: fasting glucose levels between 100 and 125 mg/dl;
  Impaired glucose tolerance: 2 hours' OGTT values between 140 and 199 mg/dl;
Time Frame: 6, 12 and 24 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Insulin Treatment for Hyperglycemia | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 15/18 | 10/18
Other Adverse Events (participants affected / at risk) | 15/18 | 14/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Treatment for Hyperglycemia (N=18) | Standard of Care (N=18)
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 8 (9)
Urinary Tract Infection (Renal and urinary disorders) | 6 (6) | 4 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Treatment for Hyperglycemia (N=18) | Standard of Care (N=18)
Abdominal Pain (Gastrointestinal disorders) | 7 (7) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 8 (8) | 6 (6)
Diarrhea (Gastrointestinal disorders) | 13 (13) | 10 (10)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (1)
Hypertension (Cardiac disorders) | 3 (3) | 7 (7)
Low Vitamin D (Endocrine disorders) | 3 (3) | 9 (9)
Nausea/Vomiting (Gastrointestinal disorders) | 8 (8) | 7 (7)

LIMITATIONS AND CAVEATS:
The original trial design was to include 250 participants. Data from the Austrian site has not been provided to the PI, thus limiting the analysis to a much smaller population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-20): https://cdn.clinicaltrials.gov/large-docs/31/NCT01683331/Prot_SAP_000.pdf